CLINICAL TRIAL: NCT02417350
Title: A Randomized Controlled Diet Intervention Comparing Effects of a Ketogenic Diet Versus a National Food Administration Recommended Diet Among Healthy Female Adults
Brief Title: Ketogenic Diet - a Randomized, Controlled, Cross-over Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: LCHF-100
Record Dates: First submitted 2015-03-27; First posted 2015-04-15 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
MeSH Terms: interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketogenic diet first (Experimental): Starting with ketogenic diet first and then switching to a NFA recommended diet
  Interventions: Other: Ketogenic diet for four weeks, then a 15 week washout, and finally a NFA recommended diet for four weeks
- NFA recommended diet first (Experimental): Starting with NFA recommended diet first and then switching to a ketogenic diet
  Interventions: Other: NFA recommended diet for four weeks, then a 15 week washout, and finally a ketogenic diet for four weeks.

INTERVENTIONS:
Other: Ketogenic diet for four weeks, then a 15 week washout, and finally a NFA recommended diet for four weeks
  Arms: Ketogenic diet first
Other: NFA recommended diet for four weeks, then a 15 week washout, and finally a ketogenic diet for four weeks.
  Arms: NFA recommended diet first

SUMMARY:
The investigators planned study is a randomized, controlled exploratory study of a ketogenic and a NFA (National Food Administration) recommended diet. Study participants will be female nutrition students with both knowledge and interest in dietary surveys, in order to increase motivation and adherence. They will be provided with cooked food. The women should be weight stable and maintain their physical activity during the study, in order to evaluate how the diet itself affects various health parameters. The investigators intend to investigate diet specific biomarkers (small molecules involved in metabolism) in the blood, as well as blood lipids, body composition, gut microbiota, energy substrate utilization, exercise performance, resting metabolic rate, hormones, cognition and sweet cravings. In addition, the investigators intend to qualitatively study the experience of following both of these dietary regimes. The investigators intend to make a short and controlled study. The study is expected to reveal whether the ketogenic diet is a healthy or unhealthy diet in the short term. The investigators also expect that data from this study will be a helpful tool to measure diet adherence in future long-term studies.

DETAILED DESCRIPTION:
Aim: The aim of this randomized controlled exploratory study is to study effects of a ketogenic diet (a low carb - high fat (LCHF) diet) compared to a National Food Administration (NFA) recommended diet (NNR2012).

Primary outcomes are blood lipids and diet specific biomarkers. Power calculations show that 20 participants are needed to obtain significant results with 90% power at the 95% significance level for the primary outcome small-dense LDL (blood lipids). The investigators calculate that 20% of the participants will drop out before the end of the study, and therefore the investigators aim to recruit a total of 24 participants.

Secondary outcomes are body composition, gut microbiota, energy substrate utilization, exercise performance, resting metabolic rate (RMR), hormones, cognition, sweet cravings, and the experience of following the two dietary regimes.

Study design: Study participants will be female nutrition students with both knowledge and interest in dietary surveys, in order to increase motivation and adherence. The women should be weight stable and maintain their physical activity during the study, in order to evaluate how the diet itself affects various health parameters.

Study participants will be provided with all food in the diet intervention. The amount and source of fat, protein and carbohydrates in the two diets are strictly defined; LCHF: Maximum 25 g carbohydrates/day (approximately 5 E%), 20 E% protein and 75 E% fat (35 E% saturated fat). NNR2012: 50 E% carbohydrates, 20 E% protein and 30 E% fat (10 E% saturated fat).

Study participants will be randomized with respect to their physical activity level to one of two study arms, with crossover design:

Study arm 1: LHCF (4 weeks) --- washout (15 weeks) --- NNR (4 weeks) Study arm 2: NNR (4 weeks) --- washout (15 weeks) --- LCHF (4 weeks)

Study participants will eat each diet for four weeks. The different diets are separated by a washout period when they eat "as usual".

Every morning during each four-week diet period the participants will measure their urine ketones by using urine ketone strips, weigh themselves and record their body weight. Any discrepancies in food intake will be recorded in a log book in which also the daily physical activity level is specified. Energy expenditure will be measured for three days during the four week periods using SenseWear activity meter (a validated and objective method) to see if energy intake matches energy expenditure.

Baseline- and outcome measurements will be performed prior to and at the end of each four-week diet period.

Qualitative measurements: When the whole diet study is completed and the research subjects have experience of eating both NNR and LCHF diet interviews will be conducted with some of the research subjects.

The study is expected to reveal whether LCHF is a healthy or unhealthy diet in the short term. The investigators also expect that data from this study will be a helpful tool to measure diet adherence in future long-term studies.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-30
* BMI 18,5-25

Exclusion Criteria:

* Waist circumference ≥80 cm
* Gravidity
* Diabetes
* Thyroid disease
* Prescribed medication for high cholesterol or high blood pressure
* Nicotine use
* Eating disorder
* Dietary restrictions

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Biomarkers in blood Measured with gaschromatography (GC)-time-of-flight/mass spectrometry (MS) and Bio-Plex Assays | baseline - four weeks
  Measured with gaschromatography (GC)-time-of-flight/mass spectrometry (MS) and Bio-Plex Assays
Blood lipids Measured with LipoPrint System | baseline - four weeks
  Measured with LipoPrint System

SECONDARY OUTCOMES:
Body composition Measured with DXA (Dual Energy X-Ray Absorptiometry) | baseline - four weeks
  Measured with DXA (Dual Energy X-Ray Absorptiometry)
Gut microbiota measured with High-throughput sequencing of nucleic acids (DNA/RNA), short-chain fatty acids | baseline - four weeks
  High-throughput sequencing of nucleic acids (DNA/RNA), short-chain fatty acids
Energy substrate utilization during submaximal exercise Measured with indirect calorimetry during ergometer cycling, lactate in blood. | baseline - four weeks
  Measured with indirect calorimetry during ergometer cycling, lactate in blood.
Exercise performance | baseline - four weeks
  Cycling at a sub-maximal work rate with increments every 4 min for three periods, thereafter increased work rate every minute until voluntary exhaustion.
Hand grip endurance | baseline - four weeks
  Hand grip test.
Resting metabolic rate Measured with indirect calorimetry | baseline - four weeks
  Measured with indirect calorimetry (Quark RMR, COSMED)
Hormones Measured with Bio-Plex Assays and ELISA | baseline - four weeks
  Measured with Bio-Plex Assays and ELISA
Cognition Measured with the Stroop color-word test | baseline - four weeks
  Measured with the Stroop color-word test
Sweet cravings Measured with a likert scale questionnaire | baseline - four weeks
  Measured with a likert scale questionnaire
Mood and appetite Measured with a likert scale questionnaire | baseline - every third day during the diet intervention period - four weeks
  Measured with a likert scale questionnaire
Experiences of following a particular dietary regime measured with Semi-structured interviews analyzed with content analysis | After finishing both study arms
  Semi-structured interviews analyzed with content analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Burén, PhD, Principal Investigator — Umeå University
Locations (1):
- Department of Food and Nutrition, Umeå, Umeå, Sweden